CLINICAL TRIAL: NCT01918709
Title: A Randomized, Open Label, Multiple Dose, Cross-over, Phase I Trial to Evaluate a Pharmacokinetic Drug Interaction and Safety Between Valsartan and Rosuvastatin in Healthy Male Volunteers
Brief Title: Drug Interaction and Safety Between Valsartan and Rosuvastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-VRCL001
Record Dates: First submitted 2013-07-22; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension, Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Valsartan 160mg, Rosuvastatin 20mg (Experimental): Both Valsartan 160mg and Rosuvastatin 20mg are administered daily by mouth once a day for 7 days.
  Interventions: Drug: Sequence 1 : Period 1(V) Period 2(R) Period 3(V+R); Drug: Sequence 2 : Period 1(V+R) Period 2(V) Period 3(R); Drug: Sequence 3 : Period 1(R) Period 2(V+R) Period 3(V); Drug: Sequence 4 : Period 1(V+R) Period 2(R) Period 3(V); Drug: Sequence 5 : Period 1(R) Period 2(V) Period 3(V+R); Drug: Sequence 6 : Period 1(V) Period 2(V+R) Period 3(R)
- Rosuvastatin 20mg (Experimental): Rosuvastatin 20mg is administered daily by mouth once a day for 7 days.
  Interventions: Drug: Sequence 1 : Period 1(V) Period 2(R) Period 3(V+R); Drug: Sequence 2 : Period 1(V+R) Period 2(V) Period 3(R); Drug: Sequence 3 : Period 1(R) Period 2(V+R) Period 3(V); Drug: Sequence 4 : Period 1(V+R) Period 2(R) Period 3(V); Drug: Sequence 5 : Period 1(R) Period 2(V) Period 3(V+R); Drug: Sequence 6 : Period 1(V) Period 2(V+R) Period 3(R)
- Valsartan 160mg (Experimental): Valsartan 160mg is administered daily by mouth once a day for 7 days.
  Interventions: Drug: Sequence 1 : Period 1(V) Period 2(R) Period 3(V+R); Drug: Sequence 2 : Period 1(V+R) Period 2(V) Period 3(R); Drug: Sequence 3 : Period 1(R) Period 2(V+R) Period 3(V); Drug: Sequence 4 : Period 1(V+R) Period 2(R) Period 3(V); Drug: Sequence 5 : Period 1(R) Period 2(V) Period 3(V+R); Drug: Sequence 6 : Period 1(V) Period 2(V+R) Period 3(R)

INTERVENTIONS:
Drug: Sequence 1 : Period 1(V) Period 2(R) Period 3(V+R) — Valsartan = Antihypertensive drug / Rosuvastatin = Antihyperlipidemic drug
  Other Names: V= Valsartan = brand name : Diovan; R= Rosuvastatin = brand name : Crestor
Drug: Sequence 2 : Period 1(V+R) Period 2(V) Period 3(R) — Valsartan = Antihypertensive drug / Rosuvastatin = Antihyperlipidemic drug
  Other Names: V= Valsartan = brand name : Diovan; R= Rosuvastatin = brand name : Crestor
Drug: Sequence 3 : Period 1(R) Period 2(V+R) Period 3(V) — Valsartan = Antihypertensive drug / Rosuvastatin = Antihyperlipidemic drug
  Other Names: V= Valsartan = brand name : Diovan; R= Rosuvastatin = brand name : Crestor
Drug: Sequence 4 : Period 1(V+R) Period 2(R) Period 3(V) — Valsartan = Antihypertensive drug / Rosuvastatin = Antihyperlipidemic drug
  Other Names: V= Valsartan = brand name : Diovan; R= Rosuvastatin = brand name : Crestor
Drug: Sequence 5 : Period 1(R) Period 2(V) Period 3(V+R) — Valsartan = Antihypertensive drug / Rosuvastatin = Antihyperlipidemic drug
  Other Names: V= Valsartan = brand name : Diovan; R= Rosuvastatin = brand name : Crestor
Drug: Sequence 6 : Period 1(V) Period 2(V+R) Period 3(R) — Valsartan = Antihypertensive drug / Rosuvastatin = Antihyperlipidemic drug
  Other Names: V= Valsartan = brand name : Diovan; R= Rosuvastatin = brand name : Crestor

SUMMARY:
Primary objective : To investigate pharmacokinetics after concomitant administration of valsartan and rosuvastatin compared to single administration of valsartan or rosuvastatin in healthy male volunteers

Secondary objective : To investigate safety profiles after the administration of valsartan or rosuvastatin alone and concomitant administration of valsartan and rosuvastatin in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male of 20 to 45 years of age at screening
2. 19 kg/m2 ≤ BMI≤ 27 kg/m2 at screening
3. 90 mmHg ≤SBP<140 mmHg and 60 mmHg ≤DBP<90 mmHg at sitting position at screening
4. At screening

   * AST and ALT ≤ 1.5 times of upper normal limit
   * Serum total bilirubin ≤ 1.5 times of upper normal limit
   * CK ≤ 2 times of upper normal limit
5. A subject who is able to understand the study, to participate whole periods of the study and to provide written informed consent voluntarily after being fully informed of the study objectives, procedures and study drug

Exclusion Criteria:

1. A subject who has medical history of or has clinically significant hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrinological, neurologic, hematologic/oncologic, or cardiovascular disease
2. A subject with severe renal insufficiency (CrCL < 10mL/min by Cockcroft-Gault estimation)
3. A subject with a history of gastrointestinal disease (e.g., ulcer, Crohn's disease) or surgery (except a simple appendectomy or repair of a hernia) that may influence the absorption of the study drug
4. A subject with a history of drug allergies to valsartan, rosuvastatin, or other drugs (e.g., aspirin, antibiotics), or a history of clinically significant allergies
5. A subject with a history of drug abuse or a positive urine drug screen for barbiturate, benzodiazepine, methamphetamine, cannabinoids, cocaine, or opiate
6. A subject who has taken any prescribed medication or herbal compounds within 14 days before the first drug administration. In addition, a subject who has taken any over-the-counter drug or vitamin supplement within 7 days before the first drug administration. (However, investigators made the final decision on the eligibility for the trial if all other conditions were satisfied)
7. A subject who has participated in any other clinical trial and received study drug within 60 days before the first drug administration
8. A subject who has donated a unit of blood or blood components within 60 days or 30 days, respectively, or received a transfusion before the first drug administration
9. A subject who has taken the drug which inhibits or induces drug metabolism such as barbital
10. A subject with unusual dietary habit which may influence on the administration, distribution, metabolism or excretion of drugs
11. A subject who consumes caffeine excessively (> 5 units/day)
12. A subject with consumes alcohol excessively (> 21 units/week, 1 unit = 10 mL of pure alcohol) or with a history of alcoholism
13. A heavy smoker ( >10 cigarettes/day)
14. A subject of positive result in serology tests (HBV, HCV, HIV, or syphilis)
15. A subject who has hereditary muscle disease or family history of hereditary muscle disease, or who has history of muscle disorder induced by drug
16. The investigator determines whether or not the subject is eligible for the study after, for example, reviewing clinical laboratory results, ECG result, or for other reason

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
PK parameters of valsartan and rosuvastatin | 0h (pre-dosing on 6d, 20d, 34d) and 0h (pre-dosing), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 16h, 24h, 48h, and 72h (on 7d, 21d, 35d). Day 1 0h (only in period 1)
  Cmax,ss and AUCτ,ss of valsartan and rosuvastatin

SECONDARY OUTCOMES:
PK parameters of valsartan and rosuvastatin | 0h (pre-dosing on 6d, 20d, 34d) and 0h (pre-dosing), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 16h, 24h, 48h, and 72h (on 7d, 21d, 35d). Day 1 0h (only in period 1)
  * Tmax,ss, Cmin,ss, t1/2,β of valsartan and rosuvastatin
  * Cmax,ss and AUCτ,ss of N-desmethyl rosuvastatin

OTHER OUTCOMES:
Safety | -1d and 1d, 2d, 3d, 4d, 5d, 6d, 7d, 8d, 9d, 10d of Period 1, 2, 3 and 42±2d
  1. Adverse event monitoring
  2. Clinical laboratory test
  3. Vital signs
  4. Electrocardiography
  5. Physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Wook Ko, Professor, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Samsung Medical Center
Locations (1):
- Clinical Trial Center, Samsung Medical Center, Seoul, South Korea